CLINICAL TRIAL: NCT05718349
Title: FGF19 in Obstructive Cholestasis: "Unveil the Signal"
Acronym: FOCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicole Hildebrand (Other)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Sponsor-Investigator, Nicole Hildebrand, Coordinating Investigator, Academisch Ziekenhuis Maastricht
Organization: Academisch Ziekenhuis Maastricht (Other)
Other Study IDs: EK172/17
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cholestasis; Icterus; Cholangiocarcinoma; Pancreatic Neoplasms; Liver Metastasis Colon Cancer
MeSH Terms: conditions — Cholestasis; Jaundice; Cholangiocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From the patients participating in the study i) blood, ii) tissue from resected material, iii) bile, iv) stool, v) urine, vi) jejunal content and vii) information on the itch severity will be collected. Since the blood vessels indicated below are easily accessible in patients undergoing pylorus-preserving pancreaticoduodenectomy (pp Whipple) or liver resection, these patients are eligible for the study and will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-cholestasis: Patients planned for pancreaticoduodenectomy or liver resection (with or without hepaticojejunostomy) who do not have cholestasis preoperatively.
  Interventions: Other: Biospecimen sampling
- Drained: Patients planned for pancreaticoduodenectomy or liver resection (with or without hepaticojejunostomy) who had cholestasis and underwent ERCP (endoscopic retrograde choledochopancreatography) with stenting to normalize the enterohepatic circulation.
  Interventions: Other: Biospecimen sampling
- Cholestasis: Patients planned for pancreaticoduodenectomy or liver resection (with or without hepaticojejunostomy) who have cholestasis preoperatively and did not undergo drainage.
  Interventions: Other: Biospecimen sampling

INTERVENTIONS:
Other: Biospecimen sampling — From the patients participating in the study i) blood, ii) tissue from resected material, iii) bile, iv) stool, v) urine, vi) jejunal content and vii) information on the itch severity will be collected.

SUMMARY:
Rationale: Bile salts are potent signalling molecules influencing various metabolic and functional processes. Bile salts exert these functions by activating nuclear (e.g. FXR ) and plasma cell membrane-bound receptors (e.g. TGR5) which are expressed in several tissues (e.g. liver, small intestine, colon, kidney and gallbladder). Bile salts regulate their own biosynthesis by controlling the transcription of the hepatic bile salt synthetic enzyme CYP7A1. Two pathways are involved in the negative feedback control of bile salt synthesis: i) the hepatic FXR-SHP pathway and ii) the ileal FXR-FGF19 pathway. Studies showed that the latter is more prominent in controlling CYP7A1 transcript levels (viz. bile salt synthesis). Thus, bile salts are synthesized in the liver, excreted in bile and expelled by the gallbladder into the proximal intestine (to aid in lipid absorption and digestion) and reabsorbed in the terminal ileum to recycle back to the liver via portal blood. Bile salts reclaimed from the intestinal lumen by the ileocyte, activate FXR. This induces the expression of an enterokine, FGF19, which signals via portal blood to the liver to activate its receptor which initiates downstream signalling to repress bile salt synthesis. The FXR/FGF19 signalling pathway is the subject of the present study.

Patients with obstructive cholestasis (=accumulation of bile) caused by malignancies (e.g. pancreatic cancer, cholangiocarcinoma) have a perturbed enterohepatic cycle. Obstructive cholestasis is associated with i) gut barrier dysfunction, ii) endotoxemia, iii) bacterial overgrowth and iv) liver injury. Previous study showed that FGF19 is expressed in the liver of patients with obstructive cholestasis. However, knowledge about the contribution of FGF19 protein by the gut in obstructive cholestasis has thus far been unexplored. Preliminary findings revealed that FGF19 is produced by the portal drained viscera (viz. intestine) of non-cholestatic patients undergoing liver surgery. The inter-organ signalling of FGF19 in an obstructed entero-hepatic cycle has not yet been characterized and likewise the metabolic and other functional effects of inflicted FGF19 signalling during cholestasis have not been clarified.

The hypothesis is that the FXR-FGF19 pathway is disturbed in patients with obstructive cholestasis, and this is associated with organ injury and metabolic dysfunction. The investigators postulate that FGF19 is not produced by the terminal ileum under conditions of obstructive cholestatic, but production is shifted to the liver and this affects metabolic processes.

The aim of this study is to investigate FGF19 signalling in patients with cholestasis compared to non-cholestatic patients or post-cholestatic patients (drained patients) by calculating fluxes across the portal drained organs. Secondly, the investigators aim to investigate the metabolic and functional consequences (glucose, lipid homeostasis, cholestatic itch, gut barrier function) of a disturbed FXR-FGF19 pathway in humans. This study will provide insights that may lead to potential therapeutic strategies for patients with a disturbed enterohepatic cycle (e.g. cholestatic liver diseases).

Study population: Adult (>18 years old) cholestatic (cholestasis group), drained (restored enterohepatic cycle) and non-cholestatic patients (controls, normal enterohepatic circulation) undergoing pancreaticoduodenectomy (Whipple procedure) for hepatopancreaticobiliary malignancies (e.g. pancreatic cancer, cholangiocarcinoma) or liver resection for hepatic malignancies (e.g. cholangiocarcinoma, colorectal liver metastases) are eligible for this study.

Study period: inclusion is planned from 1.12.2017 until 1.12.2024

DETAILED DESCRIPTION:
Because bile salts are biological emulsifiers, they play an essential role in digestion and absorption of dietary lipids and fat soluble vitamins. Bile salts also act as potent signaling molecules targeting bile salt sensing nuclear and plasma cell membrane bound receptors. Several metabolic and biological processes are influenced by activation of these receptors, including bile salt and glucose homeostasis, thermogenesis, intestinal barrier function and liver regeneration.

Bile salts are synthesized in the liver, and efficiently returned to the liver via the intestinal lumen and portal blood (enterohepatic circulation = EHC). Hepatic bile salt content is tightly regulated at multiple levels to maintain non-toxic levels. The transcription factor Farnesoid X Receptor (FXR) plays a key role in bile salt homeostasis by regulating synthesis, biliary excretion, intestinal reuptake and metabolism of bile salts. Genetic deficiency of FXR in mice results in impaired gut barrier function, dysregulated hepatic metabolism and impaired recovery from cholestatic liver injury. Bile salts repress their own biosynthesis, and this encompasses activation of FXR by bile salts in the enterohepatic tissue and controlling the transcription of Cyp7a1 in the liver (rate limiting enzyme of bile salt synthesis). Activated hepatic FXR represses the bile salt synthetic enzyme Cyp7a1 by inducing the expression of Shp. On the other hand, activated FXR in the ileum induces the expression of FGF19 which signals to the liver to repress the expression of Cyp7a1. The liver is considered to be the primary target of FGF19 as it expresses both components of the FGF19 -receptor complex (FGFR4-βklotho). Animal experiments demonstrated a crucial role of intestinal FXR in preventing bacterial overgrowth and maintaining intestinal integrity in a mouse model of obstructive cholestasis. Moreover, intestinal FXR activation ameliorated cholestatic liver injury in bile duct-ligated mice. This emphasizes that an intact EHC is crucial to maintain tissue homeostasis in the small intestine and the liver.

Intraluminal bacterial overgrowth, translocation of microbial endotoxins, increased intestinal permeability, activation of intestinal and hepatic inflammatory cascades and endotoxemia occurs frequently in patients with obstructive cholestasis (e.g. pancreatic cancer and cholangiocarcinoma). Absence of bile in the intestinal tract is associated with these anomalies. The investigators postulate that normal bile flow in patients with obstructive cholestasis is impaired and therefore bile salt signaling is impaired leading to dysregulation in enterohepatic tissues. To further improve our understanding of bile salt-FGF19 signaling across different abdominal organs, the investigators will obtain blood samples not only from the radial artery, the portal and the hepatic vein, but also from the superior mesenteric vein, inferior mesenteric vein, the splenic vein and the renal vein. By including these blood vessels, the investigators will be able to obtain information about the contribution of the small intestine, the colon, the spleen and the kidneys, separately in the production or extraction of FGF19 in humans. Namely, arteriovenous differences (ΔAV) and net organ fluxes (flow x ΔAV) serve as a quantitative measure of metabolite exchange across the portal drained viscera (PDV), the splanchnic area and the small intestine, colon, spleen and kidneys.

The hypothesis is that FGF19 inter-organ flux shifts during obstructive cholestasis towards production or release of FGF19 by other abdominal organs rather than the small intestine. Serum FGF19 elevation and FGF19 mRNA expression in the liver of patients with obstructive cholestasis support this concept.

The aim of this study is to investigate FGF19 signalling in patients with cholestasis compared to non-cholestatic patients by calculating fluxes across the portal drained organs. Secondly, the investigators will investigate the metabolic and functional consequences (glucose, lipid homeostasis, cholestatic itch, gut barrier function, bile salt composition) of a disturbed FXR-FGF19 pathway in humans. Findings from this study will provide novel insights into enterohepatic bile salt-FGF19 signaling in humans and may lead to potential therapeutic strategies in cholestatic liver diseases.

Primary objective

• Determine in vivo inter-organ fluxes of FGF19 in patients with obstructive cholestasis compared with non-cholestatic patients and drained patients

Secondary objectives

* Determine organ fluxes of bile salts (species) in patients with obstructive cholestasis compared with non-cholestatic patients (control group) and drained patients (restored EHC group)
* Determine gene expression of genes implicated in bile salt and FGF19 signaling in enterohepatic tissues (liver, jejunum, gallbladder, common bile duct, white adipose tissues), and skeletal muscle tissue of patients with obstructive cholestasis compared with non-cholestatic patients (control group) and drained patients (restored EHC group).
* Determine microbiota of patients with obstructive cholestasis compared with non-cholestatic patients (control group) and drained patients (restored EHC group) in preoperative stool and intraoperative intraluminal fecal content.
* Determine bile salt composition in patients with non-cholestatic patients (control group) and drained patients (restored EHC group) in plasma, urine and bile.
* Determine whether fluxes of metabolites (e.g. bile salts, FGF19) are related to cholestatic itch

From the patients participating in the study i) blood, ii) tissue from resected material, iii) bile, iv) stool, v) urine, vi) jejunal content and vii) information on the itch severity will be collected. Since the blood vessels indicated below are easily accessible in patients undergoing pylorus-preserving pancreaticoduodenectomy (pp Whipple) or liver resection, these patients are eligible for the study and will be included. Prior to blood sampling, the blood flow of the portal vein and hepatic artery will be measured immediately with the Transonic blood flow meter. Blood will be sampled from the following vessels:

portal vein, hepatic vein, superior mesenteric vein, inferior mesenteric vein, splenic vein, renal vein, radial artery

Arteriovenous differences (ΔAV) and net organ fluxes (flow x ΔAV) are a quantitative measure of the role of the liver, PDV, the splanchnic area, small intestine, colon, spleen and the kidneys in producing or extracting FGF19 and bile salts. The fluxes will be calculated by measuring plasma levels of metabolites and determining blood flow in these vessels.

All patients undergoing pp Whipple or liver resection have an arterial catheter during surgery from which the investigators can sample blood. The mentioned veins (6x) will be punctured directly using 25G needles. 10 ml of arterial blood and 10 ml intra-abdominal blood from the different vessels separately will be sampled once during surgery resulting in a total amount of sampled blood of maximally 70 ml. All blood samples will be collected in both pre-chilled EDTA and heparinized vacuum tubes and centrifuged at 3500 rpm at 4°C for 10 minutes. Plasma will be stored in Eppendorf cups at -80°C until further analysis. Blood flow will be measured using intra-operative Duplex ultrasonography.

Tissues will be explored by histology (histochemistry, immunohistochemistry/fluorescent), and for detailed analysis of genes implicated in bile salt-FGF19 signaling and metabolic processes (e.g. glucose homeostasis, lipid homeostasis). The following tissues (from resected material) during surgery will be collected allowing detailed study of genes implicated in bile salt-FGF19 signaling in enterohepatic tissues:

liver specimen (in case of liver resection), gallbladder specimen, common bile duct specimen, proximal jejunal specimen (in case of hepaticojejunostomy during surgical procedure), white adipose tissue (WAT) [subcutaneous, omental, visceral], rectus abdominis muscle

Previous study showed that human bile contains high levels of FGF19. However, the exact functional role of FGF19 in bile is not known. Therefore, bile will be collected intra-operatively to investigate the effect of obstructive cholestasis on FGF19 levels in bile. Bile will be collected by puncture of the gallbladder after removal or from the hepatic bile duct in case the gallbladder is not in situ.

The gut microbiota plays a major role in bile salt homeostasis by secondary modification and deconjugation of primary bile salts. The microbial composition (e.g. shift in bile salt hydrolase producing bacteria) of preoperative stool and proximal jejunal content during surgery will be analyzed. Plasma from the three patient groups (control, drained and cholestatic) will be analyzed for markers of enterocyte function (e.g. citrulline) and enterocyte damage (e.g. IFABP), transmural damage (SM22), endotoxins (LBP), pro-inflammatory cytokines (IL-6 and TNF-alpha) and novel markers for hepatic inflammation (Cathepsin).

Cholestatic pruritis (itch) is common in patients with obstructive cholestasis. The source of itch is currently unknown, and bile salts are implicated in the development of cholestatic itch. Therefore the investigators would like to ask the patients to score their itch intensity on the day before surgery by means of a Visual Analogue Scale (VAS, a scale from 0 (no itch) to 10 (worst itch possible)). In addition, the investigators will ask them to fill in a short questionnaire, the 5D itch scale. Metabolites implicated in itch (e.g. bile salts) will be analyzed in the blood samples to calculate fluxes and these will be correlated with the preoperative VAS scores and 5D itch scale.

Urine will also be collected preoperatively of all patients to investigate whether cholestasis influences the route of bile salt excretion (from biliary excretion to renal excretion). Bile salt composition will be analyzed in urine with liquid chromatography mass spectrometry (LC-MS).

Main study parameters/endpoints: The main study parameter is the net organ flux of FGF19 across abdominal organs calculated by measuring FGF19 levels in human plasma using an enzyme-linked immuno-sorbent assay (ELISA) in cholestatic versus non-cholestatic patients and drained patients. Human plasma will be obtained during surgery from 7 vessels i) radial artery, ii) mesenteric superior vein, iii) mesenteric inferior vein, iv) renal vein, v) splenic vein, vi) hepatic vein and vii) portal vein to calculate net organ fluxes. Secondary parameters are expression of genes related to bile salt and FGF19 signaling in enterohepatic tissues (liver, jejunum, gallbladder, common bile duct, white adipose tissue and skeletal muscle tissue), genes implicated in glucose and lipid homeostasis, FGF19 levels in bile, gut microbiota, cholestatic itch and bile salt composition in urine.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients planned for a Whipple procedure or liver resection are included. Informed consent will be obtained either at the outpatient ward or at the day of admission, with one week time to decide. Patients will then also have time to ask questions.

Blood from these patients will be sampled during surgery under general anesthesia from the portal vein, hepatic vein, superior mesenteric vein, inferior mesenteric vein, splenic vein, renal vein and the radial artery. The experimental set-up consists of 1 time arterial blood sampling (10ml) and 1 time intra-abdominal blood sampling (6x10ml) which is maximal 70 ml in total. During surgery blood flow will be measured of the portal vein and hepatic artery to precisely calculate organ fluxes. The portal vein and hepatic artery are easy accessible for flow measurement with the Transonic flow meter. This device is CE-certified and used routinely to measure actual blood flow. No risks are associated with measuring of these blood flows.

Additionally, bile will be sampled during surgery (4 ml) from the gallbladder or hepatic duct during surgery, and biopsies will be taken from the liver (1, in case of liver resection), gallbladder (1), jejunum (1, in case of hepaticojejunostomy), common bile duct (CBD, 1). white adipose tissue (WAT, from three sites; subcutaneous, omental and visceral adipose tissue) and rectus abdominis muscle for gene expression studies of genes. Moreover, perioperative stool and urine, and jejunal content during surgery (in case of hepaticojejunostomy) will be collected for detailed analysis of microbiota/bile salt composition to investigate the effect of obstructive cholestasis on these parameters. Patients will be assessed for severity of itch by a questionnaire (visual analog scale and 5D itch scale) on the day before surgery to correlate fluxes to cholestatic itch.

The methods applied, i.e. arterial and intra-abdominal blood sampling and collecting liver/jejunal biopsies as part of planned resection, have been used previously without any consequences for the surgical procedures or the patients. In comparison to previously ethical approved protocols, bile (4 ml) will be sampled from the gallbladder or hepatic duct during surgery, and biopsies of the gallbladder (1x), CBD (1x) and WAT (3x), as well as stool will be collected one time preoperatively. There are no additional risks related to the collection of bile and tissues since these are part of the resected tissues. The biopsy of the small intestine, white adipose tissue, and rectus abdominis muscle will be taken from parts that will be resected during the surgery or from the surgical incision site, thus preventing the risk for permanent complications. Potential peroperative bleeding of the tissue will be electrocoagulated by the surgeon. Abdominal biopsies will be taken by skilled hepatopancreaticobiliary surgeons. No further risk is associated with the collection of preoperative stool and urine. Although the results of this project have no direct positive effects for the patients involved, they do contribute to the understanding of the role of bile salts and FGF19 signaling under cholestatic conditions. Insights from this study would provide novelty and substantial knowledge in possible effects of FGF19 therapy in cholestatic liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pp Whipple or liver resection
* Age >18 and <75 years

Exclusion Criteria:

* Jejunostomy
* Lactation, pregnancy and planning of pregnancy
* Inflammatory bowel disease
* Alcohol or drug abuse within 1 year
* Inborn errors of bile salt synthesis
* Failure to give informed consent or refusal to store patient data for fifteen years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive jaundice undergoing pp Whipple or liver resection are eligible for this study. Controls are non-jaundiced and drained patients undergoing pp Whipple or liver resection. The rationale for including patients undergoing pp Whipple or liver resection is that the nature of the surgical procedure in the abdomen allows sampling of blood from the portal drained organs, and tissue sampling. Patients will be recruited at the surgical outpatient clinic of Maastricht University Medical Center (MUMC+) and University Hospital RWTH Aachen (Germany). Patients in the cholestasis group (group III), will be included largely at the University Hospital RWTH Aachen. Ten to twenty percent of the cholestasis group can be included in MUMC+.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
plasma FGF19 levels | Intraoperatively
  A factor which signals to the liver to repress the expression of Cyp7a1 (rate limiting enzyme of bile salt synthesis)
plasma bile salt levels | Intraoperatively
  Bile salts are synthesized in the liver, and efficiently returned to the liver via the intestinal lumen and portal blood
Gene expression levels of genes implicated in bile salt homeostasis and FGF19 signaling | Intraoperatively
  in liver, proximal jejunum, gallbladder, common bile duct, subcutaneous adipose tissue, omental adipose tissue, visceral adipose tissue, and rectus abdominis muscle
Biliary FGF19 level | Intraoperatively
  A factor which signals to the liver to repress the expression of Cyp7a1 (rate limiting enzyme of bile salt synthesis)
itch intensity | Preoperatively
  by means of a Visual Analogue Scale (VAS, a scale from 0 (no itch) to 10 (worst itch possible))
Enterocyte damage | Intraoperatively
  Plasma IFABP
Enterocyte function | Intraoperatively
  Plasma Citrulline
Transmural intestinal damage | Intraoperatively
  Plasma SM22
Endotoxinemia | Intraoperatively
  Plasma LBP
Bile salt composition | Preoperatively
  In stool, jejunal content, plasma, and urine
Bile salt composition | Intraoperatively
  In stool, jejunal content, plasma, and urine
Microbial composition | Preoperatively
  In stool and jejunal content
Microbial composition | Intraoperatively
  In stool and jejunal content

CONTACTS AND LOCATIONS:
Overall Officials: Steven Olde Damink, MD, PhD, Principal Investigator — Academisch Ziekenhuis Maastricht
Locations (1):
- RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hofmann AF. The enterohepatic circulation of bile acids in mammals: form and functions. Front Biosci (Landmark Ed). 2009 Jan 1;14(7):2584-98. doi: 10.2741/3399. PMID 19273221
- [Background] Schaap FG, Trauner M, Jansen PL. Bile acid receptors as targets for drug development. Nat Rev Gastroenterol Hepatol. 2014 Jan;11(1):55-67. doi: 10.1038/nrgastro.2013.151. Epub 2013 Aug 27. PMID 23982684
- [Background] McEwan HP. Treatment of severe toxaemia of pregnancy. Lancet. 1972 Feb 12;1(7746):374. doi: 10.1016/s0140-6736(72)92862-0. No abstract available. PMID 4109754
- [Background] Modica S, Petruzzelli M, Bellafante E, Murzilli S, Salvatore L, Celli N, Di Tullio G, Palasciano G, Moustafa T, Halilbasic E, Trauner M, Moschetta A. Selective activation of nuclear bile acid receptor FXR in the intestine protects mice against cholestasis. Gastroenterology. 2012 Feb;142(2):355-65.e1-4. doi: 10.1053/j.gastro.2011.10.028. Epub 2011 Nov 2. PMID 22057115
- [Background] Goodwin B, Jones SA, Price RR, Watson MA, McKee DD, Moore LB, Galardi C, Wilson JG, Lewis MC, Roth ME, Maloney PR, Willson TM, Kliewer SA. A regulatory cascade of the nuclear receptors FXR, SHP-1, and LRH-1 represses bile acid biosynthesis. Mol Cell. 2000 Sep;6(3):517-26. doi: 10.1016/s1097-2765(00)00051-4. PMID 11030332
- [Background] Xie MH, Holcomb I, Deuel B, Dowd P, Huang A, Vagts A, Foster J, Liang J, Brush J, Gu Q, Hillan K, Goddard A, Gurney AL. FGF-19, a novel fibroblast growth factor with unique specificity for FGFR4. Cytokine. 1999 Oct;11(10):729-35. doi: 10.1006/cyto.1999.0485. PMID 10525310
- [Background] Hart RA, Woo SL, Newton PO. Ultrastructural morphometry of anterior cruciate and medial collateral ligaments: an experimental study in rabbits. J Orthop Res. 1992 Jan;10(1):96-103. doi: 10.1002/jor.1100100112. PMID 1727939
- [Background] Parks RW, Clements WD, Smye MG, Pope C, Rowlands BJ, Diamond T. Intestinal barrier dysfunction in clinical and experimental obstructive jaundice and its reversal by internal biliary drainage. Br J Surg. 1996 Oct;83(10):1345-9. doi: 10.1002/bjs.1800831007. PMID 8944448
- [Background] Wells CL, Jechorek RP, Erlandsen SL. Inhibitory effect of bile on bacterial invasion of enterocytes: possible mechanism for increased translocation associated with obstructive jaundice. Crit Care Med. 1995 Feb;23(2):301-7. doi: 10.1097/00003246-199502000-00016. PMID 7867356
- [Background] Bloemen JG, Venema K, van de Poll MC, Olde Damink SW, Buurman WA, Dejong CH. Short chain fatty acids exchange across the gut and liver in humans measured at surgery. Clin Nutr. 2009 Dec;28(6):657-61. doi: 10.1016/j.clnu.2009.05.011. Epub 2009 Jun 11. PMID 19523724
- [Background] Schaap FG, van der Gaag NA, Gouma DJ, Jansen PL. High expression of the bile salt-homeostatic hormone fibroblast growth factor 19 in the liver of patients with extrahepatic cholestasis. Hepatology. 2009 Apr;49(4):1228-35. doi: 10.1002/hep.22771. PMID 19185005
- [Background] Zweers SJ, Booij KA, Komuta M, Roskams T, Gouma DJ, Jansen PL, Schaap FG. The human gallbladder secretes fibroblast growth factor 19 into bile: towards defining the role of fibroblast growth factor 19 in the enterobiliary tract. Hepatology. 2012 Feb;55(2):575-83. doi: 10.1002/hep.24702. Epub 2011 Dec 19. PMID 21953282
- [Background] Mraz M, Lacinova Z, Kavalkova P, Haluzikova D, Trachta P, Drapalova J, Hanusova V, Haluzik M. Serum concentrations of fibroblast growth factor 19 in patients with obesity and type 2 diabetes mellitus: the influence of acute hyperinsulinemia, very-low calorie diet and PPAR-alpha agonist treatment. Physiol Res. 2011;60(4):627-36. doi: 10.33549/physiolres.932099. Epub 2011 May 16. PMID 21574752
- [Background] Galman C, Angelin B, Rudling M. Pronounced variation in bile acid synthesis in humans is related to gender, hypertriglyceridaemia and circulating levels of fibroblast growth factor 19. J Intern Med. 2011 Dec;270(6):580-8. doi: 10.1111/j.1365-2796.2011.02466.x. Epub 2011 Nov 2. PMID 22003820
- [Background] Kuipers F, Bloks VW, Groen AK. Beyond intestinal soap--bile acids in metabolic control. Nat Rev Endocrinol. 2014 Aug;10(8):488-98. doi: 10.1038/nrendo.2014.60. Epub 2014 May 13. PMID 24821328
- [Background] Schreuder TC, Marsman HA, Lenicek M, van Werven JR, Nederveen AJ, Jansen PL, Schaap FG. The hepatic response to FGF19 is impaired in patients with nonalcoholic fatty liver disease and insulin resistance. Am J Physiol Gastrointest Liver Physiol. 2010 Mar;298(3):G440-5. doi: 10.1152/ajpgi.00322.2009. Epub 2010 Jan 21. PMID 20093562